CLINICAL TRIAL: NCT04515030
Title: Changes of Trace Elements in Aqueous Humor, Blood and Tears of Patients With Primary Glaucoma and Analysis of Related Factors
Brief Title: Changes of Trace Elements in Aqueous Humor, Blood and Tears and Analysis of Related Factors
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020KYPJ120
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2021-12

CONDITIONS: Primary Glaucoma
Keywords: trace element; Age-related cataract; Aqueous humor, blood, tears.; Flow-Injection-Inductively-Coupled-Plasma-Mass-Spectrometry; Metabonomics; Genomics
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor, blood, tears.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary glaucoma: Primary glaucoma patients were diagnosed based on guidelines [1-2]. Patients with a confirmed diagnosis of primary glaucoma were enrolled and classified into the acute angle-closure crisis (AACC), primary angle-closure glaucoma (PACG), and primary open-angle glaucoma (POAG) subgroups.
  1. Prum BE, Herndon LW, Moroi SE, et al. Primary Angle Closure Preferred Practice Pattern® Guidelines. Ophthalmology 2016;123:P1-40. doi:10.1016/j.ophtha.2015.10.049
  2. Prum BE, Rosenberg LF, Gedde SJ, et al. Primary Open-Angle Glaucoma Preferred Practice Pattern® Guidelines. Ophthalmology 2016;123:P41-111. doi:10.1016/j.ophtha.2015.10.053
- Senile cataract: Senile cataract patients were diagnosed based on guideline [3]. Patients with a confirmed diagnosis of senile cataract were enrolled and considered as controls for aqueous humor-related analysis.
  [3] Olson RJ, Braga-Mele R, Chen SH, et al. Cataract in the Adult Eye Preferred Practice Pattern®. Ophthalmology 2017;124:P1-119. doi:10.1016/j.ophtha.2016.09.027
- Normal control: Normal people without ocular diseases were enrolled as normal control.

SUMMARY:
Trace elements are one of the indispensable substances in human body and play an important physiological role. Zinc is a trace element second only to iron in organisms, which is widely distributed in various systems and organs and plays an important biological role, and interacts with other trace elements such as copper and iron. With the improvement of detection methods, it is possible to detect the concentration of zinc and other trace elements in liquid samples. It is reported in the existing literature that there are significant changes in the concentration of trace elements in a variety of eye diseases. Our group intends to collect three kinds of samples (aqueous humor, blood and tears) of patients with primary glaucoma and age-related cataract who were treated in Sun Yat-sen Eye Center of Sun Yat-sen University from March 2020 to March 2021. Normal people with matched age and sex were recruited as normal control group (normal control group only collected blood and tear samples). Three methods (FI-ICP-MS, metabonomics and genomics) were used to study the concentration changes of patients with primary glaucoma in three kinds of body fluid samples, and the related factors were analyzed combined with clinical data, so as to provide a theoretical basis for studying the pathogenic mechanism and new prevention pathway of primary glaucoma.

DETAILED DESCRIPTION:
Glaucoma is a group of optic nerve diseases characterized by progressive and irreversible degeneration of retinal ganglion cells and their axons. There are different opinions on the pathogenesis of glaucoma, which further reflects that the mechanism of glaucoma optic nerve injury is still in the exploratory stage, and there is still a long way to go to develop effective drugs to prevent or reverse the visual function damage in patients with glaucoma. Therefore, on the basis of previous studies, our research group explored and expanded whether there were similar pathological changes in patients with clinical glaucoma not only in aqueous humor, but also in blood and tear samples, and further studied the mechanism. Three kinds of samples (aqueous humor, blood and tears) were collected from patients with primary glaucoma and age-related cataract treated in Sun Yat-sen Eye Center of Sun Yat-sen University. Normal people with matched age and sex were recruited as normal control group (normal control group only collected blood and tear samples). Three methods of inductively coupled plasma mass spectrometry (FI-ICP-MS), metabonomics and genomics were used to study the concentration changes of patients with primary glaucoma in three kinds of body fluid samples, and the related factors were analyzed combined with clinical data, so as to provide a new theoretical basis for studying the pathogenic mechanism and new prevention pathway of primary glaucoma.

ELIGIBILITY:
Inclusion Criteria:

- If you meet the following conditions, you can participate in our study and become a subject in the case group:

1. those who are over 50 years old and can complete all the examinations and examinations.
2. other secondary and developmental factors have been excluded and diagnosed as primary glaucoma.
3. before anti-glaucoma surgery, you can take part in blood sampling examination and collect sufficient tears, and sufficient aqueous humor can be collected during the operation.

If you meet the following conditions, you can participate in our study and become a subject in the disease control group:

1. those who are over 18 years old and can complete all the tests and examinations.
2. other factors have been excluded and age-related cataract has been clearly diagnosed.
3. before cataract surgery, you can take part in blood sampling examination and collect sufficient tears, and sufficient aqueous humor can be collected during the operation.

If you meet the following conditions, you can participate in our study and become a normal control group:

1. those who are over 50 years old and can complete all the tests and examinations.
2. No previous history of ophthalmopathy (except ametropia, strabismus and age-related cataract).
3. normal eye examination (intraocular pressure < 21mmHg, chamber angle open, cup / plate ratio normal, visual field normal).
4. can cooperate with those who take part in blood test and collect enough tears. -

Exclusion criteria:

1. those who have a history of eye trauma, eye surgery or eye laser.
2. elevated intraocular pressure and glaucoma optic nerve damage caused by secondary or developmental factors (such as neovascularization, uveitis, trauma, lens-related factors, surgery, drugs, etc.).
3. suffering from other eye diseases that may affect metabolism (such as uveitis, ocular neovascularization, age-related macular degeneration, etc.) and major systemic diseases (such as heart disease, hypertension, hyperlipidemia, diabetes, hepatitis, digestive tract malabsorption, hypothyroidism, vitamin deficiency, mental illness, severe psoriasis, malignant tumors, etc.).
4. pregnant, lactating and pregnant women.
5. those who refuse to sign the informed consent form due to discomfort or other reasons or voluntarily withdraw from the researcher.
6. those who are unable to cooperate with the relevant inspection and inspection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary glaucoma. Age-related cataract. Normal population.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
The concentrations of trace elements in aqueous humor, blood, and tears. | Specimens were collected before and after surgery for approximately 1 years.
  The aqueous humor, blood, and tears samples were collected from patients with primary glaucoma, senile cataract, and normal people. The concentrations of trace elements were measured by inductively coupled plasma mass spectrometry (FI-ICP-MS), metabonomics and genomics.

CONTACTS AND LOCATIONS:
Overall Officials: Yiqing Li, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University, China
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weinreb RN, Khaw PT. Primary open-angle glaucoma. Lancet. 2004 May 22;363(9422):1711-20. doi: 10.1016/S0140-6736(04)16257-0. PMID 15158634
- [Background] Li Y, Andereggen L, Yuki K, Omura K, Yin Y, Gilbert HY, Erdogan B, Asdourian MS, Shrock C, de Lima S, Apfel UP, Zhuo Y, Hershfinkel M, Lippard SJ, Rosenberg PA, Benowitz L. Mobile zinc increases rapidly in the retina after optic nerve injury and regulates ganglion cell survival and optic nerve regeneration. Proc Natl Acad Sci U S A. 2017 Jan 10;114(2):E209-E218. doi: 10.1073/pnas.1616811114. Epub 2017 Jan 3. PMID 28049831
- See also: Primary Open-Angle Glaucoma — https://pubmed.ncbi.nlm.nih.gov/15158634/
- See also: Mobile Zinc Increases Rapidly in the Retina After Optic Nerve Injury and Regulates Ganglion Cell Survival and Optic Nerve Regeneration — https://pubmed.ncbi.nlm.nih.gov/28049831/